

| Study Title | Dual-Task Zumba Gold for Improving the Cognition of<br>Community-Dwelling Older Adults With Mild Cognitive<br>Impairment: A Pilot Randomized Controlled Trial |
|---|---|
| <b>Document Description</b> | Information Sheet and Consent |
| <b>Document Date</b> | February 08, 2021 |
| NCT Number | Pending |



#### INFORMATION SHEET

# Dual-Task Zumba Gold for Improving the Cognition of Community-Dwelling Older Adults With Mild Cognitive Impairment: A Pilot Randomized Controlled Trial

We would like to invite you to participate in this study. Before you decide to take part, it is important for you to understand why the research is being done and what will it involve. Please take time to read the following information and feel free to ask any questions.

# Purpose of the study

This study aims to determine the feasibility and preliminary efficacy of an intervention to promote physical and cognitive training for community-dwelling older adults with mild cognitive impairment. This will be done by using Zumba Gold dance with integrated cognitive exercises, which aims to enhance cognitive function of older adults at risk for dementia.

#### **Invitation of potential participants**

Taking part in the research in purely voluntary. This study will include persons aged 55 or above with mild cognitive impairment (with subjective cognitive complaints and validated by objective screening tools to be administered). Those with uncontrolled medical conditions that would limit the program safety and regularly taking medications that could influence cognitive function will not be invited to participate.

#### **Involvement of the participants**

Once you agree to participate, baseline data will be gathered which include demographic data, health history, cognitive function, mood, quality of life, physical mobility, and bodily measures (e.g., weight, height, waist circumference, blood pressure).

Participants will be randomly allotted into two groups: (1) dual-task Zumba Gold (DTZ) group or (2) health education group. The activity in the first group will involve Zumba Gold dance enriched with cognitive exercises, to be done 3x per week for 60 minutes, for a duration of 12 weeks. The sessions will include basic and low-impact steps which are tailor-made for older people. It will be conducted as a group (of 10 participants) at the community gym and will be facilitated by a licensed Zumba Gold dance instructor and project assistants. Alternatively, participants in the second group will receive health education about dementia risk reduction through physical and mental activities.

After the program's completion in 12 weeks, you will be asked to rate its feasibility and acceptability through a short survey. Some participants may be requested for an interview to gather feedback and suggestions to help improve the activity. Measures assessed before the start of the program will be evaluated after its 12<sup>th</sup> week, with a follow-up assessment after 6 weeks.

# Benefits and risks in participation

Participation in this project could potentially promote various health benefits such as improving your physical activity, psychosocial status, and cognitive function. Eventually, this study could support the development of programs and future studies which will improve dementia risk reduction services for community-based older adults.

Risks may be involved, as you may need to provide information that you may find personal, but rest assured that they will remain confidential and will never be shared with any non-member of the research team. Since this will involve a physical activity program, you may experience fatigue during the activity. To prevent such, rest periods every 10–15 minutes and light refreshments will be provided in

between and after the activity. Your vital signs will also be monitored before, during, and after the activity to ascertain your safety. In case of any untoward events such as chest pain, dizziness, or falls, appropriate medical attention and first aid will be provided. The investigators will shoulder necessary medical fees for any untoward event attributed to the study.

# **Confidentiality of information**

It is an important responsibility of the research team to keep all the information confidential. Instead of your name, control numbers will be used to maintain your anonymity. Moreover, the results of the study will be presented without any personal identifiers. Only members of the research team that will have access to the documents of the study.

#### Results of the study

The results of the study will be combined and analyzed anonymously. The researcher may contact you for purposes of clarification in the information provided, as needed. The written report will also be submitted for publication in a peer-reviewed journal. You will not have any identifiable information from any published material.

#### **Review of the study procedures**

The study plan has been reviewed by the Institutional Review Board of the Hong Kong Polytechnic University (HSESC Reference Number: ). They have assessed that the study meets the requirement for scientific ethical conduct.

## Rights of the participants

You have every right to withdraw from the study, before or during the program, without penalty of any kind. You also have the right to request access to the data you have provided for this project. If you would like further information about this study, please contact Dr Angela Leung at angela.ym.leung@polyu.edu.hk. If you have any complaints about the conduct of this study, you may contact the Human Subjects Ethics Sub-Committee of The Hong Kong Polytechnic University (c/o Research Office of the University), clearly stating the responsible person and department of this study as well as the HSESC Reference Number.

Thank you for your interest in participating in this study.



# CONSENT TO PARTICIPATE

| Ι, | , consent to p | articipate | e in the focus | group i | nterview | as part of |
|---|---|---|---|---|---|---|
| the study entitled: Dual-Task<br>Dwelling Older Adults With M | Zumba Gold | for Imp | roving the Co | ognitio | n of Co | nmunity- |
| Trial. | | | | | | |
| (Please check ✓ the following b | ooxes to indica | te unders | tanding) | | | |
| ☐ The procedure as set out in the | ne attached info | ormation | sheet has bee | n fully | explaine | d. |
| □ I understand the benefits and | risks involved | l. | | | | |
| <ul> <li>My participation in the proje<br/>of any kind.</li> </ul> | ct is voluntary | and I car | n withdraw at | any tin | ne withou | ıt penalty |
| ☐ I have also been given the answered clearly. | opportunity to | ask que | estions about | the stu | dy and h | ave been |
| ☐ I understand that information However, my right to privacy w | | | | - | | |
| ☐ I acknowledge that I have the researcher anytime. | right to questi | ion any p | art of the proc | edure a | nd can co | ontact the |
| ☐ I understand that if I have contact participant, I may contact angela.ym.leung@polyu.edu.hk | ct: Mobile | | | | | |
| Participant's Signature: | | | | ate: | / | _/ |
| Researcher's Signature: | | | | ate: | / | _/ |
| Witness' Name/Signature: | | | Γ | ate: | / | / |